CLINICAL TRIAL: NCT05644275
Title: MechBRACE - The Influence of Demographic Parameters and ACL Injury on the Association Among Clinical, Functional and Biomechanical Parameters
Brief Title: The Influence of Demographic Parameters and ACL Injury on the Association Among Clinical, Functional and Biomechanical Parameters
Acronym: MechBRACE
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-01851; mu22Egloff
Record Dates: First submitted 2022-11-30; First posted 2022-12-09 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Anterior Cruciate Ligament (ACL) Injury
Keywords: limb symmetry index (LSI); muscle strength; single leg hop (SLH) distance; Leg symmetry index for SLH (LSISLH distance)
MeSH Terms: conditions — Wounds and Injuries | interventions — Data Collection; Demography; Functional Status

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Data collection (demographic, clinical, functional and biomechanical outcomes in patients after ACL injury (conservative therapy and/or surgery) in patients of different ages and healthy controls) — Analysis of existing data from previous research projects MechSens (EKNZ 2019-01315) and RetroBRACE I and II (EKNZ 2019-00491 and EKNZ 2020-00551) as descriptive statistics (mean, standard deviation, range) for all parameters (for female or male patients with ACL injury and healthy subjects).

SUMMARY:
This retrospective study aims at analysing demographics and clinical, functional and biomechanical outcomes in patients after ACL injury (conservative therapy and/or surgery) in patients of different ages and healthy controls. Demographics, as well as clinical, functional and biomechanical parameters were collected between 2019 and 2022 in two research projects approved by the Ethikkommission Nordwestschweiz (EKNZ 2019-00491, EKNZ 2019-01315, EKNZ 2020-00551). The primary research question analyzes if maximal SLH distance and LSISLH distance are related to the predictors age, sex, isokinetic muscle strength and the presence of injury.

DETAILED DESCRIPTION:
Injury of the anterior cruciate ligament (ACL) is one of the most common injuries of the knee. ACL reconstruction using auto- and allografts is still the gold-standard technique and widely used in the surgical treatment of ACL ruptures. Potential deficits in the affected leg are frequently evaluated using the limb symmetry index (LSI) calculated as performance affected side/performance unaffected side x 100. Several factors other than injury may influence single leg hop (SLH) distance and LSI such as sex, age, and muscle strength. This retrospective study aims at analysing demographics and clinical, functional and biomechanical outcomes in patients after ACL injury (conservative therapy and/or surgery) in patients of different ages and healthy controls. Demographics, as well as clinical, functional and biomechanical parameters were collected between 2019 and 2022 in two research projects approved by the Ethikkommission Nordwestschweiz (EKNZ 2019-00491, EKNZ 2019-01315, EKNZ 2020-00551)

ELIGIBILITY:
Inclusion Criteria:

* Patients: 2-10 years since ACL injury
* Control subjects: no previous injury to the meniscus or the ligament apparatus of the knee

Exclusion Criteria:

* Bilateral injury or previous injury or surgical treatment of the opposite side within the past 2 years and the injured leg within the past 6 months
* Concomitant conditions that affect the mobility of the knee (e.g., neuromuscular diseases that affect lower limb movement, injury of the posterior cruciate ligament (PCL), more than one collateral ligament ruptured, fracture, luxation of the knee, tumorous disease, immunosuppressed patients)
* Inability to give informed consent

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All parameters of patients after ACL injuries and healthy controls assessed in the Laboratory for Functional Biomechanics, University Hospital Basel in two prior projects will be included in this study. All data were collected in research projects that had ethical approval and participants signed informed consent forms for the respective research project:
  * Comparison between augmented ACL repair and ACL reconstruction (RetroBRACE, EKNZ 2019-00491 and RetroBRACE II, EKNZ 2020-00551)
  * Evaluating the relationship of in vivo ambulatory load and mechanosensitive cartilage biomarkers (MechSens, EKNZ 2019-01315)
Sampling Method: Non-Probability Sample
Enrollment: 181 (Actual)
Dates: Start 2022-11-02 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Peak value for SLH distance | one time assessment at baseline
  Peak value for SLH distance (for female or male patients with ACL injury and healthy subjects). This test is to jump as far as possible on a single leg, without losing balance and landing firmly. The distance is measured from the start line to the heel of the landing leg. The goal is to have a less than 10% difference in hop distance between the injured limb and uninjured limb.
Leg symmetry index for SLH (LSISLH distance) | one time assessment at baseline
  Leg symmetry index for SLH (LSISLH distance) for healthy (non-dominant/dominant side*100) and for ACL injured (ACL injured/contralateral*100). Leg symmetry index (LSI) calculated as performance affected side/performance unaffected side x 100. A commonly regarded threshold for the LSI is 90%, corresponding to a 10% deficit, which is considered physiological.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Egloff, PD Dr. med., Principal Investigator — University Hospital Basel, Clinic for Orthopedics and Traumatology
Locations (1):
- University Hospital Basel, Orthopedics and Traumatology, Basel, Switzerland